CLINICAL TRIAL: NCT04882592
Title: Noninvasive Spinal Neuromodulation Enables Locomotor Recovery in Individuals With Cerebral Palsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SpineX Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SPNX-00
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Therapeutic Arm (Experimental): Spinal Cord Neuromodulation with SCiP during Activity Based NeuroRehab Therapy
  Interventions: Device: SCiP
- Sham Arm (Sham Comparator): Sham Stimulation during Activity Based NeuroRehab Therapy
  Interventions: Device: SCiP

INTERVENTIONS:
Device: SCiP — Noninvasive spinal cord neuromodulator

SUMMARY:
Assessing the effects of noninvasive spinal cord neuromodulation on improving function in individuals with cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* 1) individuals above the age of 2 years of age and 2) diagnosed with cerebral palsy (CP). The exclusion criteria included 1) children with selective dorsal root rhizotomy, 2) intramuscular Botox injection in the preceding 12 months, 3) current antispastic medications 4) unhealed fractures or contractures that would prevent them from performing functional tasks and 5) tendon lengthening surgeries.

Exclusion Criteria:

* Intramuscular Botox injection in the past 12 months

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Stepping overground or on a treadmill | 3 months
Gross Motor Functional Measure (GMFM) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- SpineX, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hastings S, Zhong H, Feinstein R, Zelczer G, Mitrovich C, Gad P, Edgerton VR. A pilot study combining noninvasive spinal neuromodulation and activity-based neurorehabilitation therapy in children with cerebral palsy. Nat Commun. 2022 Oct 5;13(1):5660. doi: 10.1038/s41467-022-33208-w. PMID 36198701